CLINICAL TRIAL: NCT01914497
Title: Dipole Density Right Atrial Mapping and Assessment of Therapy In Cavotricuspid Isthmus Flutter
Brief Title: Dipole Density Mapping of Typical Atrial Flutter
Acronym: DDRAMATIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acutus Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CL-AFL-002
Record Dates: First submitted 2013-07-31; First posted 2013-08-02 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Atrial Flutter
MeSH Terms: conditions — Atrial Flutter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acutus Medical System (Experimental): Proprietary software algorithms will be used generate electrical activation maps based dipole density data acquired by the Acutus Medical Catheter during the procedures. These activation maps will then be applied to a 3D model of the endocardial surface to create a 3D activation map.
  Interventions: Device: Acutus Medical System Mapping

INTERVENTIONS:
Device: Acutus Medical System Mapping

SUMMARY:
Study to determine the feasibility of the Acutus Medical System in obtaining data to create Dipole Density Maps of electrical activation in the right atrium in patients with typical atrial flutter.

ELIGIBILITY:
Inclusion Criteria:

1. Be aged 18 to 75 years
2. Be scheduled for ablation of typical atrial flutter (cavotricuspid isthmus dependent)
3. Be able and willing to give informed consent

Exclusion Criteria:

1. Have any of the following:

   1.1 Patients with implanted prosthetic, artificial, or repaired cardiac valves in the chamber being mapped.

   1.2 Patients with permanent pacemaker or ICD leads in the chamber being mapped. 1.3Patients with hypercoagulopathy or an inability to tolerate anticoagulation therapy during an electrophysiology procedure.
2. Require treatment in the left atrium and/or a require a transseptal puncture to access the left atrium during the index procedure
3. Have had a myocardial infarction within the prior two months
4. Have had cardiac surgery within the prior three months
5. Have an intracardiac thrombus
6. Have clinically significant tricuspid valve regurgitation or stenosis
7. Have had any cerebral ischemic event (including transient ischemic attacks) in the prior six months
8. Be pregnant or nursing
9. Be currently enrolled in any other clinical investigation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Incidence of device-and procedure-related adverse events | 7 days
The number of patients in which offline construction of pre- and post-treatment activation maps can be completed | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Willems, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Germany